CLINICAL TRIAL: NCT00174707
Title: A Phase III Randomized Study of Sequential Epidoxorubicin Followed By CMF: Cyclophosphamide+Methotrexate+Fluorouracil (Arm A) Versus Sequential Epidoxorubicin Followed By Docetaxel Followed By CMF (Arm B) Versus Sequential Intensified Epidoxorubicin Followed By Docetaxel Followed By High-Dose Cyclophosphamide (Arm C) in Early Breast Cancer Patients With Positive Axillary Lymph Nodes
Brief Title: Study of Docetaxel in Breast Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Medical Director, Sanofi-aventis aministrative office
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAX_IT1_302; TAX_IT_216
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Methotrexate; Docetaxel; Cyclophosphamide

ARMS (3):
- A (Active Comparator): Sequential Epidoxorubicin followed by CMF: ciclophosphamide/Methotrexate/fluorouracile (±TAM: tamoxifen)
  Interventions: Drug: epidoxorubicine, ciclophosphamide, methotrexate, fluorouracile
- B (Experimental): Sequential Epidoxorubicin followed by Docetaxel followed by ciclophosphamide/methotrexate/fluorouracile (± TAM)
  Interventions: Drug: epidoxorubicine, docetaxel, ciclophosphamide, methotrexate, fluorouracile
- C (Experimental): Sequential Intensified Epidoxorubicin followed by Docetaxel followed by Cyclophosphamide (± TAM)
  Interventions: Drug: epidoxorubicine, docetaxel, cyclophosphamide

INTERVENTIONS:
Drug: epidoxorubicine, ciclophosphamide, methotrexate, fluorouracile — Sequential Epidoxorubicin followed by ciclophosphamide/Methotrexate/fluorouracile (±TAM)
  Arms: A
Drug: epidoxorubicine, docetaxel, ciclophosphamide, methotrexate, fluorouracile — Sequential Epidoxorubicin followed by Docetaxel followed by ciclophosphamide/methotrexate/fluorouracile (± TAM)
  Arms: B
Drug: epidoxorubicine, docetaxel, cyclophosphamide — Sequential Intensified Epidoxorubicin followed by Docetaxel followed by Cyclophosphamide (± TAM)
  Arms: C

SUMMARY:
Primary objectives:

* To compare the disease free survival (DFS) in patients treated with the sequential epidoxorubicin, cyclophosphamide, methotrexate, and fluorouracil (CMF) regimen to that in patients treated with the same treatment plus docetaxel given sequentially after epidoxorubicin

Secondary objectives:

* To compare the DFS in patients treated with the sequential epidoxorubicin, docetaxel and CMF (only patients with > or = 4 lymph nodes) regimen to that in patients treated with sequential intensified epidoxorubicin/docetaxel/high dose (HD) cyclophosphamide regimen
* To evaluate the overall survival in each arm
* To evaluate the tolerability of a sequential intensified epidoxorubicin/docetaxel/HD-cyclophosphamide (arm C)
* To compare the safety of a sequential epidoxorubicin/docetaxel/CMF (arm B) regimen versus a standard sequential epidoxorubicin/CMF regimen (arm A)

ELIGIBILITY:
Inclusion criteria:

* Histologically proven breast cancer at the first diagnosis with > or = 4 axillary nodes showing evidence of tumor among a minimum of 10 resected lymph nodes (American Joint Committee on Cancer 1992 pathologic staging pT1-4, pN1-2 [at least 1/10], M0)
* Ages ≥ 18 years and ≤ 70 years for patients who will be randomized to arm A and B. Ages ≥ 18 years and ≤ 65 years for patients who will be randomized to arm C
* World Health Organization performance status 0-1
* Definitive surgical treatment must be either mastectomy or breast conserving surgery, with axillary lymph node dissection for operable breast cancer (clinical T1-3, N1, M0). Margins of resected specimen from definitive surgery must be histologically free of invasive adenocarcinoma and ductal carcinoma in situ. Lobular carcinoma in situ does not count as a positive margin. Patients with histologically-documented infiltration of the skin (pT4a) will be also eligible
* Surgical procedures completed within 8 weeks from the randomization.
* Laboratory requirements:

  * Hematology :

    * Neutrophils ≥ 2 x 10^9/L
    * Platelets ≥ 100 x 10^9/L
    * Hemoglobin ≥ 10 g/DL
  * Hepatic function:

    * Total bilirubin ≤ 1 time the upper-normal limits of the institutional normal values.
    * ASAT & ALAT ≤ 2.5 UNL, alkaline phosphatase ≤ 5 UNL. Patients with ASAT &/or ALAT > 1.5 x UNL associated with alkaline phosphatase > 2.5 x UNL are not eligible for the study
  * Renal function :

    * Creatinine ≤ 140 µmol/L (1.6 mg/DL); if limit values, the creatinine clearance should be performed and should be ≥ 60 ml/min
* Normal left ventricular ejection fraction or superior to the lower limits of the institution
* Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating center
* Complete work-up within 3 months prior to randomization. All patients will have bilateral mammography, chest X rays (posteroanterior [PA] and lateral), abdominal ultrasound and/or computed tomography scan, & bone scan

Exclusion criteria:

* Axillary lymph nodes free of involvement
* Primary breast cancer with histology other than adenocarcinoma
* Inflammatory carcinoma
* Any locally advanced (T4 and/or N2-known N3) or metastatic (M1) breast cancer
* Past or current history of ipsilateral or contralateral invasive or contralateral ductal in situ breast carcinoma. A past or current history of ipsilateral ductal in situ or lobular in situ (ipsilateral or contralateral) breast carcinoma is not an exclusion criterion
* Histologically positive resection margins. Patients undergoing conservative resection margins can be considered eligible if radically resected within 4 weeks from randomization
* Pregnant or lactating women or women of childbearing potential (e.g. not using adequate contraception)
* History of prior or concomitant malignancies other than curatively treated basal cell skin cancer or excised cervical carcinoma in situ
* Symptomatic peripheral neuropathy > grade 2 according to the National Cancer Institute Common Toxicity Criteria
* Other serious illnesses or medical conditions:

  * Congestive heart failure or angina pectoris even if it is medically controlled. Previous history of myocardial infarction within 1 year from study entry, uncontrolled high risk hypertension or arrhythmias
  * History of significant neurologic or psychiatric disorders including dementia or seizures
  * Active infection
  * Peptic ulcer, unstable diabetes mellitus or other contraindications for the use of dexamethasone
* Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational regimen within 30 days prior to study entry
* Concurrent treatment with any other anti-cancer therapy
* Concurrent treatment with ovarian hormonal replacement therapy. Prior treatment should be stopped before study entry
* Prior systemic anticancer therapy for breast cancer (chemotherapy, hormonal therapy, immunotherapy, etc.) as adjuvant and/or neo-adjuvant therapy
* Concomitant treatment with corticosteroids used for reasons other than premedication; however, patients receiving chronic treatment with corticosteroids (>6 months) at low dose (≤ 20 mg of methylprednisolone or equivalent dose of other corticosteroids) for whichever reason are eligible
* Definite contraindications for the use of corticosteroids as premedication
* Prior radiation therapy

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 998 (Actual)
Dates: Start 1997-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Invasive Disease-Free Survival (IDFS) - with exclusion of ductal carcinoma in situ- DCIS- either collateral or ipsilateral, according to STEEP in adjuvant breast cancer trial: Standardized Definitions for Efficacy Endpoints | Time between randomization date and date of local or distant recurrence or contralateral breast cancer or second primary (non breast) cancer or death from any cause, whichever occurs first

SECONDARY OUTCOMES:
Recurrence-Free Survival (RFS) | Time between the date of randomization and the date of local or distant recurrence or death from any cause, whichever occurs first, thus excluding contralateral breast cancer or second primary (non breast) cancers
Overall Survival (OS) | Time between the date of randomization and date of death
Distant Disease-Free Survival (DDFS) | Time betwen the date of randomization and the date of distant recurrence or death from any cause, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Georges Paizis, MD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Milan, Italy